CLINICAL TRIAL: NCT03095144
Title: A Retrospective Comparative Study, Post Operative Outcomes of Pyloromyotomy Procedure Under Spinal Anesthesia Compared to General Anesthesia
Brief Title: Spinal Anesthesia and General Anesthesia for Pyloromyotomy - Surgical Outcomes a Comparison Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MOSTAFA.SOMRI, DIRECTOR OF ANESTHESIA DEPARTEMT, Bnai Zion Medical Center
Other Study IDs: BnaiZionMC-17-MS-001
Record Dates: First submitted 2017-03-19; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Hypertrophic Pyloric Stenosis; Spinal Anesthesia; General Anesthesia
Keywords: pyloromyotomy; spinal anaesthesia; surgical outcomes; general anaesthesia; infants
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Spinal anesthesia: Lumbar puncture was performed with a midline approach through either the fourth or fifth lumbar space using a 22 or 25 -gauge 4 cm disposable styletted needle. Spinal isobaric Bupivacaine 0.5%, 0.8-1 mg.kg-1 without epinephrine was injected using a 1ml tuberculin syringe.
  Interventions: Device: Spinal anesthesia
- General anesthesia: The General anesthesia is preformed by intravenous Propofol (2-4 mg.kg-1) and Fentanyl (1-2 µg.kg-1) and Rocuronium bromide (0.5mg.kg-1) administration to facilitate endotracheal intubation, assisted by Sellick manoeuvre. Anaesthesia maintenance with Sevoflurane (2-3%) in an air/oxygen mixture, intravenous Fentanyl as required.
  Interventions: Device: General anesthesia

INTERVENTIONS:
Device: Spinal anesthesia — Pyloromyotomy under spinal anesthesia
  Groups: Spinal anesthesia
Device: General anesthesia — Pyloromyotomy under general anesthesia
  Groups: General anesthesia

SUMMARY:
Background: The purpose of this retrospective study is to evaluate surgical outcomes of pyloromyotomy in infants performed under spinal anesthesia compares to general anesthesia.

Methods: After receiving the approval of the hospital ethics committee, retrieving, reviewing files and collecting data. Primary outcomes: total operating room time, duration of surgery, pain management and postoperative apnea episodes, time of regaining full enteral feeding. Secondary outcome measures: include cardio-respiratory changes and events, and substantial vomiting postoperatively.

DETAILED DESCRIPTION:
After receiving of the approval of the MedicalCenter Ethics Committee, the files of all infants with hypertrophic pyloric stenosis, who were treated by open pyloromyotomy under Spinal Anesthesia and general anesthesia in Bnai-Zion Medical Center through a decade will be reviewed.

Primary outcomes: total operation time, pain assessment and management, postoperative apnea episodes and time for regaining full enteral feeding. Secondary outcome measures include, significant cardiorespiratory changes and substantial postoperative vomiting.

Full enteral feeding is defined as an infant tolerating 130 ml.kg-1 of formula a day, or breast feeding in 6-8 divided doses. Infants tolerating 2-3 full enteral feedings without complications were discharged.

Total operating room time defined as the elapsing time since entrance to the operating room until transport to the post anesthesia care unit or neonatal intensive care unit .

Surgical time is defined as the elapsing time since performing the surgical incision until wound dressing .

All infants assisted by the CRIES pain score for pain measurement and management after surgery. The CRIES score, (which is the abbreviation of C - Crying, R - Requires increase oxygen administration, I - Increased vital signs, E - Expression, S- Sleeplessness), obtained by nurses each 4 hours.

Anesthesia pharmacological Paracetamol 25 mg.kg-1 administered rectally to all infants prior to surgery. Fentanyl 1mg.Kg-1 ordered IV by the anesthetist in titration dose for pain control in PACU, and Paracetamol 15 mg.kg-1 ordered by the paediatric surgeon rectally for postoperative pain in the surgical ward, as needed. Bilateral ultra sound- guided rectus sheath block performed at the end of surgery.

Respiratory monitoring f performed in the NICU using Vitalmon® 5010 (Kontron Instruments, France), with the nursing staff recording occurrences of apnea, desaturation, and bradycardia.

A long apnea defined as a respiratory pause of 15 seconds or longer, or any apnea that coincided with the appearance of bradycardia.

The General anesthesia is preformed by intravenous Propofol (2-4 mg.kg-1) and Fentanyl (1-2 µg.kg-1) and Rocuronium bromide (0.5mg.kg-1) administration to facilitate endotracheal intubation, assisted by Sellick manoeuvre. Anaesthesia maintenance with Sevoflurane (2-3%) in an air/oxygen mixture, intravenous Fentanyl as required.

All spinal blocks performed by the same consultant anesthesiologist group. The infant's back prepared scrubbed with chlorhexidine solution. Lumbar puncture performed with a midline approach through either the fourth or fifth lumbar space using a 22 or 25 -gauge 4 cm disposable styletted needle. Spinal isobaric Bupivacaine 0.5%, 0.8-1 mg.kg-1 without epinephrine injected using a 1ml tuberculin syringe.

Standard monitoring during anaesthesia included: heart rate, blood pressure by non-invasive means, skin temperature and blood oxygen saturation (SpO2) using the AS/3® monitor (Datex, Engestrom, Helsinki, Finland). The above monitored parameters were applied before performing the spinal block, and subsequently every 5 minutes after the spinal block, until the end of surgery. In all infants, the stomach was suctioned until no further gastric fluid was obtained.

Effective spinal block was defined by the infant's inability to move the lower extremities. The sensory level of anesthesia was determined by observing the patient's segmental response to a tetanic stimulus of 10-30 milli-amperes, delivered by a peripheral nerve stimulator (Innervator® NS252, Fisher and Pajkel Healthcare Electronics Ltd, Auckland, New Zealand). Attainment of sensory block was indicated by the lack of crying, flexure of the upper extremities and an increase in both the heart and respiratory rate by 15% above baseline.

Bradycardia is defined as less than 100 bpm, and hypoxia is defined as O2 saturation of less than 95 % for more than 30 seconds. An increase in blood pressure and heart rate of more than 15% above the baseline considered clinically significant.

All the surgical pyloromyotomy procedures were performed by the same paediatric surgeon group, using open Fredet-Ramstedt technique through a supraumbilical transverse right upper quadrant incision. For inadequate relaxation or if persistent discomfort was noticed, infants who were given a single dose bolus of IV Diprivan, (0.5-1 mg.kg-1), or a titration dose of midazolam (0.05-0.1 mg.kg-1).

Intra-operatively, the infants were hydrated with 5% dextrose in a 0.45% NaCl solution at a rate of 5 ml.kg-1.h-1 using an infusion pump.

Statistical analysis:

For the demographic continuous variables (age, weight and height at surgery) and the surgical continuous variables (duration of surgery, duration of spinal anesthesia, total time in operating room, regain of full feeding time and home discharge day) means, standard deviations, medians, ranges and IQR (the difference between Q3 and Q1) will be calculated.

For the categorical variables (number of spinal attempts and sedation required), numbers and percentages will be calculated.

For the continuous repeated measures of respiratory rate, oxygen saturation rates, mean blood pressure and heart rate at six periods of times, the means and standard deviations were calculated, and the results analyzed by the Anova repeated-measures test.

All statistical tests analyzed to a significance level of 0.05. Statistical analysis performed using the STATA 12.0 software.

ELIGIBILITY:
Inclusion Criteria:

Children well hydrated: a normal serum electrolyte count;

Exclusion Criteria:

Children who's spinal puncture was unsuccessful even after a third attempt.

Ages: 4 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with HPS, treated by open pyloromyotomy under Spinal Anesthesia in our medical center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Total operating room time | 1 hour
  The elapsing time since entrance to the operating room until transport to the post anaesthesia care unit or neonatal intensive care unit in mins.
Pain management | 1-24 hours
  The CRIES score, (which is the abbreviation of C - Crying, R - Requires increase oxygen administration, I - Increased vital signs, E - Expression, S- Sleeplessness), obtained by nurses each 4 hours
Time of regaining full enteral feeding | up to 48 hours
  Time of regaining full enteral feeding

SECONDARY OUTCOMES:
Number of substantial vomiting | up to 24 hours
  Follow-up of number of vomiting events

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Somri, Prof, Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Undecided